CLINICAL TRIAL: NCT05863104
Title: An Open-label, Uncontrolled, Multicenter Study to Evaluate the Safety, Local Tolerability, Systemic Exposure, and Efficacy of 1% Glycopyrronium Bromide (GPB) Cream in Adolescents With Severe Primary Axillary Hyperhidrosis
Brief Title: Assessment of Safety, Tolerability, Systemic Exposure and Efficacy of GPB Cream in Adolescents With Severe Primary Hyperhidrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. August Wolff GmbH & Co. KG Arzneimittel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GPBK-08/2018
Record Dates: First submitted 2023-04-27; First posted 2023-05-17 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Primary Axillary Hyperhidrosis
Keywords: Excessive sweating
MeSH Terms: conditions — Hyperhidrosis | interventions — Glycopyrrolate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glycopyrronium Bromide (GPB) Cream (Experimental): Formulation containing Glycopyrronium Bromide (GPB) for topical application
  Interventions: Drug: Glycopyrronium Bromide (GPB) Cream

INTERVENTIONS:
Drug: Glycopyrronium Bromide (GPB) Cream — Application of cream to each axilla

SUMMARY:
The aim of this study is to evaluate the safety, tolerability and systemic exposure (in a subset of patients) of topical administration of 1% GPB in adolescents with severe primary axillary hyperhidrosis.

ELIGIBILITY:
Inclusion Criteria:

* Medical diagnosis of severe primary axillary hyperhidrosis with a PRHS score of ≥5 with symptoms for at least 3 months before Screening
* At least 50 mg of sweat production in each axilla measured gravimetrically over a period of 5 minutes at room temperature along with a humidity consistent with the normal climate in that area (patients have to acclimatize to that room for at least 30 minutes before the measurement)
* Adolescents of both sexes aged 12 to 17 years (until study completion) with a body mass index percentile ≥10 and ≤90 (according to Kromeyer-Hauschild et al 2001)
* Local tolerability assessment (skin reaction) score = 0

Exclusion Criteria:

* Secondary hyperhidrosis, ie, hyperhidrosis that is secondary to other underlying diseases such as (but not limited to) hyperthyroidism, lymphoma, and malaria
* Previous surgical treatment of hyperhidrosis including sympathectomy, surgical debulking of the sweat glands, subcutaneous tissue curettage, ultrasonic surgery, microwave treatment (miraDry), or laser treatment
* Botulinum toxin treatment for the treatment of axillary hyperhidrosis in the previous 4 months
* Hypersensitivity to glycopyrrolate, or to any of the excipients of the investigational medicinal product (IMP)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2023-03-07 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2024-03-06 (Actual)

PRIMARY OUTCOMES:
Number of patients with Adverse Drug Reaction during treatment | Baseline to Day 57
Number of patients with a local tolerability assessment (skin reaction score) >0 during treatment | Baseline to Day 57
Αbsolute change in GP plasma concentration from Baseline to Day 15 | Baseline to Day 15

SECONDARY OUTCOMES:
Absolute change in logarithmic values of total sweat production assessed by GM from Baseline to Day 29 | Baseline to Day 29
Absolute change in logarithmic values of total sweat production assessed by GM from Baseline to Day 57 | Baseline to Day 57
Absolute change in logarithmic values of total sweat production assessed by GM from Day 29 to Day 57 | Day 29 to Day 57
Relative change in total sweat production assessed by GM from Baseline to Day 29 and Day 57 | Baseline to Day 29 and Day 57
Relative change in total sweat production assessed by GM from Day 29 to Day 57 | Day 29 to Day 57
Proportion of responders assessed by GM at Day 29 and Day 57 | Day 29 and Day 57
Absolute change in patient-rated hyperhidrosis severity (PRHS) score from Baseline to Day 29 and Day 57 | Baseline to Day 29 and Day 57
  The patient-rated hyperhidrosis severity (PRHS) score will be assessed by asking the following question: "How did you perceive your underarm sweating in the past 24 hours? Please rate it on a scale from 0 (no sweating at all) to 10 (worst sweating that you ever had)"
Absolute change in patient-rated hyperhidrosis severity (PRHS) score from Day 29 to Day 57 | Day 29 to Day 57
  The patient-rated hyperhidrosis severity (PRHS) score will be assessed by asking the following question: "How did you perceive your underarm sweating in the past 24 hours? Please rate it on a scale from 0 (no sweating at all) to 10 (worst sweating that you ever had)"
Absolute change in the Children's dermatology life quality index (CDLQI) score from Baseline to Day 29 and Day 57 | Baseline to Day 29 and Day 57
  The Children's dermatology life quality index (CDLQI) is a simple 10-question questionnaire that assesses the burden of hyperhidrosis. It is validated for children aged 5-16 years. The answers to the questions are generally scored on a 4-point scale: 'very much' = 3, 'quite a lot' = 2, 'only a little' = 1, 'not at all' or question unanswered = 0.
  The CDLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more impairment of the child's life is experienced.
Absolute change in the Children's dermatology life quality index (CDLQI) score from Day 29 to Day 57 | Day 29 to Day 57
  The Children's dermatology life quality index (CDLQI) is a simple 10-question questionnaire that assesses the burden of hyperhidrosis. It is validated for children aged 5-16 years. The answers to the questions are generally scored on a 4-point scale: 'very much' = 3, 'quite a lot' = 2, 'only a little' = 1, 'not at all' or question unanswered = 0.
  The CDLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more impairment of the child's life is experienced.
Absolute change in GP plasma concentration from Baseline to Day 8 | Baseline to Day 8
Absolute change in GP plasma concentration from Day 8 to Day 15 | Day 8 to Day 15
Frequency, severity, and relation of ADRs, SAEs, TEAEs, SUSARs, and discontinuations due to TEAEs | Screening to 14 Days after End of Treatment
Local tolerability based on the skin reaction score | Day 1, Day 29, Day 57/End of Treatment and 14 Days after Day 57/End of Treatment
  Local tolerability at the application sites will be assessed and evaluated by the investigator using a skin reaction score: 'No evidence of irritation' = 0, 'Minimal erythema, barely perceptible' = 1, 'Definite erythema, readily visible; minimal edema or minimal popular response' = 2, 'Erythema and papules' = 3, 'Definite edema' = 4, 'Erythema, edema, and papules' = 5, 'Vesicular eruption' = 6, 'Strong reaction spreading beyond test site' = 7, 'Folliculitis' = 8.
Neurological assessment of anticholinergic effects by a 4-point scale | 7 to 4 Days before Baseline, Day 15, Day 29, Day 43, Day 57/End of Treatment
  The occurrence of possible anticholinergic effects including dry mouth, dry eyes, blurred vision, red eyes, constipation, micturition disorder, drowsiness, and concentration difficulties is rated on a 4-point scale: 'severe intensity' = 3, 'moderate intensity' = 2, 'mild intensity' = 1, 'no evidence' = 0.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Rolf-Markus Szeimies, Principal Investigator — Klinikum Vest GmbH, Knappschaftskrankenhaus Recklinghausen
Locations (1):
- Dr. Michael Sebastian, Mahlow, Germany